CLINICAL TRIAL: NCT01796444
Title: A Prospective Randomized Multicenter Phase III Study of Axillary Lymph Node Dissection Versus no Dissection in Breast Cancer With Positive Sentinel Lymph Node--the Validation of Z0011 in China
Brief Title: Axillary Lymph Node Dissection Versus no Dissection in Breast Cancer With Positive Sentinel Lymph Node
Acronym: Z0011-China
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director, Head of Breast Cancer Center, Principal Investigator, Clinical Professor, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z0011-China
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Sentinel Lymph Node Biopsy; Axillary Lymph Node Dissection
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Axillary Lymph Node Dissection (Active Comparator): After sentinel lymph node biopsy, surgery for standard axillary lymph node dissection. Pathological evaluation (include intraoperative pathological examination) is performed routinely. All women were to receive whole-breast opposing tangential-field radiation therapy. Adjuvant systemic therapy was determined by the treating physician.
  Interventions: Procedure: Sentinel Lymph Node Biopsy; Procedure: Intraoperative Pathological Examination; Procedure: Axillary Lymph Node Dissection; Procedure: Pathological Evaluation; Drug: Adjuvant Systemic Therapy; Radiation: Radiation Therapy
- Non-Axillary Lymph Node Dissection (Experimental): After sentinel lymph node biopsy, no surgery of axillary lymph node In this study, the absence of surgery is the experimental arm (non-inferiority trial). Pathological evaluation (include intraoperative pathological examination) is performed routinely. All women were to receive whole-breast opposing tangential-field radiation therapy. Adjuvant systemic therapy was determined by the treating physician.
  Interventions: Procedure: Sentinel Lymph Node Biopsy; Procedure: Intraoperative Pathological Examination; Procedure: Pathological Evaluation; Drug: Adjuvant Systemic Therapy; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy — Sentinel lymph nodes are identified with the combining use of intraoperative gamma detector and/or blue dye.
  Other Names: SLNB
Procedure: Intraoperative Pathological Examination — touch imprint cytology and/or frozen section and/or OSNA
Procedure: Axillary Lymph Node Dissection — Axillary lymph node dissection involving removal of at least level I and II nodes.
  Other Names: ALND
  Arms: Axillary Lymph Node Dissection
Procedure: Pathological Evaluation — H&E and IHC
Drug: Adjuvant Systemic Therapy — Adjuvant systemic therapy was determined by the treating physician according to the recently NCCN.
  Other Names: chemotherapy or hormone therapy
Radiation: Radiation Therapy — Whole-breast opposing tangential-field radiation therapy.

SUMMARY:
The recently randomized trial (ASCOG Z0011) support that among patients with limited sentinel lymph node (SLN) metastatic breast cancer treated with breast conservation and systemic therapy, the use of sentinel lymph node biopsy (SLNB) alone compared with axillary lymph node dissection (ALND) did not result in inferior survival. These patients, therefore, are unlikely to benefit from further surgery that results in a longer period of hospitalization, higher costs and higher postoperative morbidity. This result has been written in the 2012 National Comprehensive Cancer Network Clinical Practice Guidelines.

However, Limitations of Z0011, such as failure to achieve target accrual and possible randomization imbalance favoring the SLNB-alone group, must be considered. In the other hand, further testing in different country are needed.

The investigators design and begin a prospective randomized multicenter phase III study of ALND vs. no ALND in breast Cancer with positive SLN--the validation of Z0011 in China.

DETAILED DESCRIPTION:
OBJECTIVES:

To determine the effects of complete axillary lymph node dissection (ALND) on survival of patients with sentinel lymph node (SLN) metastasis of breast cancer.

OUTLINE: This is a randomized multicenter study. Before randomization, all women were stratified according to age (≤50 years, >50 years), tumor size(≤2cm, >2cm) and research center. All the patients underwent lumpectomy and sentinel lymph node biopsy (SLNB). Eligible women were randomly assigned to ALND or no ALND Active Comparator: Patients undergo axillary lymph node dissection involving removal of at least level I and II nodes.

Experimental: No surgery of axillary lymph node in this arm. All the patients were to receive whole-breast opposing tangential-field radiation therapy. The use of adjuvant systemic therapy was determined by the treating physician according to the recently NCCN.

Patients are followed up every 4 months for the first 2 years, every 6 months from the third year to the fifth year, and then annually for a total of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Patient aged 18 years and above;
* Patient with histological proven invasive breast cancer;
* Clinical T1-T2 disease with no distant metastasis;
* Patient with clinical N0 status;
* Patient for whom conservative surgery with sentinel lymph node (SLN) technique is feasible from the start in terms of carcinologic;
* Patient with positive SLNs 1~2;
* Signed consent to participate.

Exclusion Criteria:

* History of neoadjuvant chemotherapy or hormone therapy;
* History of breast cancer (ipsilateral, i.e. recurrence, or contralateral breast);
* History of any other invasive cancer;
* Initial metastatic disease known;
* Pregnant women or lactating women;
* Impossibility to undergo medical examinations of the study for geographical, social or psychological reasons.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | Time to relapse or progression up to 10 years
  Time from randomization to relapse or death.

SECONDARY OUTCOMES:
Overall Survival | Time to death up to 10 years
  Time from randomization to date of death.
Axillary Recurrence Rate | Time to local relapse up to 10 years
  Estimate the incidence of axillary recurrence after surgery followed by axillary dissection or after surgery alone.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-sheng Wang, MD, Study Chair — Shandong Cancer Hospital and Institute; Tao Ouyang, MD, Principal Investigator — Beijing Cancer Hospital and Institute; Jiong Wu, MD, Principal Investigator — Fudan University; Feng-xi Su, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Hong-yuan Li, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China